CLINICAL TRIAL: NCT01910831
Title: Randomized, Double-Blind, Contralateral, Controlled Study to Assess the Efficacy of DerMend Moisturizing Bruise Formula in Improving the Appearance of Chronically Aged Mature Skin of the Forearms and Hands
Brief Title: Study to Assess DerMend Moisturizing Bruise Formula in Improving the Appearance of Chronically Aged Forearms and Hands
Acronym: CCCR-28-2013
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Center for Clinical and Cosmetic Research (Other)
Collaborators: Ferndale Laboratories, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Steven Nestor, M.D., Ph.D., Director, The Center for Clinical and Cosmetic Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCCR 28-2013
Record Dates: First submitted 2013-07-25; First posted 2013-07-30 (Estimated); Results first posted 2015-04-16 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Purpura
Keywords: bruising, reduction, older age, aging
MeSH Terms: conditions — Purpura; Contusions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DerMend Moisturizing Bruise Formula (Experimental): Apply LEFT treatment to LEFT arm or (vica versa) RIGHT treatment to RIGHT arm. Will not be known to the subject which arm is on the active treatment and which is on the placebo control. Applied twice daily for 12 weeks. Each subject will have one arm/hand that is either a)the experimental treatment or b) the placebo control.
  Interventions: Drug: DerMend Moisturizing Bruise Formula
- Non-active placebo control (Placebo Comparator): Apply LEFT treatment to LEFT arm or (vica versa) RIGHT treatment to RIGHT arm. Will not be known to the subject which arm is on the active treatment and which is on the placebo control. Each subject will have one arm/hand that is either a)the experimental treatment or b) the placebo control.
  Interventions: Drug: Non-active placebo control

INTERVENTIONS:
Drug: DerMend Moisturizing Bruise Formula — DerMend Moisturizing Bruise Formula, a skin care cream containing a proprietary blend of retinol, ceramides, arnica oil, and alpha hydroxy acids and other ingredients.
  Other Names: DerMend
  Arms: DerMend Moisturizing Bruise Formula
Drug: Non-active placebo control — Non-active placebo control
  Arms: Non-active placebo control

SUMMARY:
To determine the efficacy (measured at 12 weeks) of DerMend Moisturizing Bruise Formula in improving the appearance of bruising and reducing the appearance of photoaging of the forearms and hands in mature skin. Assessments will be made through ongoing objective measurements and clinical ratings.

To confirm the safety (local tolerance) of DerMend Moisturizing Bruise Formula.

DETAILED DESCRIPTION:
Twenty subjects with mature skin, at one study center, with bruising and moderate to severe photodamage will be selected for the study. Twenty subjects will be enrolled to achieve a total of 40 arms to be analyzed. At baseline, the Subject will be instructed to use the study cream on one forearm and hand while a control cream will be used on the other. Both the study cream and the control cream will be provided in containers labeled Left and Right so that the subjects are blinded. Each cream labeled Left and Right will be randomized with either the treatment or control cream in the Left container and the opposite cream will be assigned to the Right container. Each subject will always get the control cream in one container and the treatment cream in the other container. Each subject will be randomized to apply cream Right to the right forearm and hand. Subject will apply cream Left to the left forearm and hand. At each visit, the Evaluator will count the total number of bruises, determine the size of each bruise and assess each forearm and hand for surface roughness, laxity and mottled hyperpigmentation. Furthermore, subjective investigator and subject global assessments of bruising, skin roughness, wrinkling and pigmentation will be measured. Subjects will be evaluated at weeks 0 (baseline), 2, 4, 6, 8, 10, and 12. Additionally, standardized, high-resolution digital photographs will be taken at each visit using the Vectra software..

The following scales will be used for grading these features: Roughness (degree of scaling and surface texture) - very smooth (1), mostly smooth (2), slightly rough (3), rough (4), very rough (5). Laxity (ability to spring back after pinching the skin) - very tight (1), somewhat tight (2), somewhat loose (3), loose (4), very loose (5). Mottled hyperpigmentation (a combination of lentigines and hyperpigmented and hypopigmented spots) - very even (1), mostly even with few blotches (2), blotchy (3), mostly blotchy (4), very blotchy (5).

Secondary endpoints will be measured including the speed of healing (measured by the two week average percentage change in bruising) and a reduction in the Investigator's and Subject's Global Assessment compared to baseline after twelve weeks. The following 5-point scale will be used for both the Investigator's and Subject's Global Assessments: 0, no improvement; 1, <25% improvement; 2, 25% to 50% improvement; 3, 51% to 75% improvement; and 4, >75% improvement.

Finally, adverse events, including but not limited to redness, swelling, blistering, ulceration, bleeding, itch or pain, will be monitored at each visit and assessed by both the Subject and the Evaluator.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria are eligible for this study:

1. Male and female subjects who are 60-80 years of age, with phototypes I to IV.
2. Subjects who have provided written, informed consent.
3. Subjects with multiple bruises on both forearms and hands.
4. Subjects with moderate to severe photodamage on forearms and hands.
5. Subjects with relatively equal photodamage on both forearms and hands.
6. Subjects who are willing to follow the treatment schedule.
7. Subjects who are willing to maintain their usual sunscreen or use of photoprotective clothing during outdoor activities.

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for this study:

1. Participation in a clinical drug or device research study within 30 days of enrollment or participation in a research study concurrent with this study;
2. Subjects with history of bleeding disorders;
3. Subjects with use of isotretinoin in the past 12 months;
4. Subjects with a pacemaker or internal defibrillator;
5. Subjects who take more than 2 anticoagulant therapies.
6. Treatment of any type of cancer within the last 6 months;
7. Subjects who are unable to communicate or cooperate with the Investigator due to language problems, poor mental development, or impaired cerebral function;
8. History of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure, including known sensitivities to any ingredient;
9. Concomitant use of potentially irritating over-the-counter products that contain ingredients such as arnica, alpha-hydroxy acid, salicylic acid, retinol or glycolic acid;
10. Subjects who present with one or more conditions which, in the opinion of the investigator, making the subject unsuitable for participation.
11. Subjects who apply any topicals other than the study treatment or their usual sunscreen.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nestor, MD, PhD, Principal Investigator — Director; Brian Berman, MD, PhD, Study Chair — Co-director; Julie A Santos, PA-C, CRC, Study Chair — Study Coordinator; Andrew C Frisina, MS, Study Chair — Study Coordinator
Locations (1):
- Center for Clinical and Cosmetic Research, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: DerMend — https://www.dermend.com/
- See also: Ferndale Pharma Group — http://www.ferndalepharmagroup.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment in this study is defined as follows:
  20 individual subjects were recruited to participate in the study.
  40 arms (1 left arm and 1 right arm) were analyzed for the results. The N for data analysis is "40".
Groups:
- DerMend Moisturizing Bruise Formula vs. Vehicle Control: Apply LEFT treatment to LEFT arm or (vica versa) RIGHT treatment to RIGHT arm. Will not be known to the subject which arm is on the active treatment and which is on the placebo control. Each subject will have one arm/hand that is either a)the experimental treatment or b) the placebo control.
  DerMend Moisturizing Bruise Formula vs. Vehicle control.
Period: Overall Study
Arm/Group | DerMend Moisturizing Bruise Formula vs. Vehicle Control
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: 20 Subjects were enrolled into the study. 40 arms were analyzed.
Groups:
- All Participants: Apply LEFT treatment to LEFT arm or (vica versa) RIGHT treatment to RIGHT arm. Will not be known to the subject which arm is on the active treatment and which is on the placebo control. Applied twice daily for 12 weeks. Each subject will have one arm/hand that is either a)the experimental treatment or b) the placebo control.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.60 (5.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Bruising
Description: To determine the efficacy (measured at 12 weeks) of DerMend Moisturizing Bruise Formula in improving the appearance of bruising and reducing the appearance of photoaging of the forearms and hands in mature skin.
Time Frame: 12 weeks
Population: 20 subjects were enrolled into the study in a 1:1 ratio (DerMend: Placebo Control). 40 arms were used in the final data analysis. After 84 days of treatment, there was no change in serious AEs, or any AEs. 40 arms were used in the final data analysis.
Measure: Mean (Standard Deviation); unit: cm squared
Groups:
- LEFT Arm Randomized to DerMend Moisturizing Bruise Formula: Apply LEFT treatment to LEFT arm or (vica versa) RIGHT treatment to RIGHT arm. Will not be known to the subject which arm is on the active treatment and which is on the placebo control. Applied twice daily for 12 weeks. Each subject will have one arm/hand that is either a)the experimental treatment or b) the placebo control.
  DerMend Moisturizing Bruise Formula
- LEFT Arm Randomized to Non-active Placebo Control: Apply LEFT treatment to LEFT arm or (vica versa) RIGHT treatment to RIGHT arm. Will not be known to the subject which arm is on the active treatment and which is on the placebo control. Each subject will have one arm/hand that is either a)the experimental treatment or b) the placebo control.
Arm/Group | LEFT Arm Randomized to DerMend Moisturizing Bruise Formula | LEFT Arm Randomized to Non-active Placebo Control
Number analyzed (Participants) | 20 | 20
cm squared | 3.74 (3.39) | 4.50 (3.22)

2. Secondary Outcome: Investigator Global Assessment (IGA)
Description: To determine efficacy with respect to the IGA of improving the appearance of "bruising" and reducing the appearance of photoaging of the forearms and hands:
  IGA:
  0=No improvement
  1. <25% improvement
  2. 25% to 50% improvement
  3. 51% to 75% improvement
  4. >75% improvement
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LEFT Arm Randomized to DerMend Moisturizing Bruise Formula | LEFT Arm Randomized to Non-active Placebo Control
Number analyzed (Participants) | 20 | 20
units on a scale | 1.60 (1.23) | 2.05 (1.19)

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No